CLINICAL TRIAL: NCT05693155
Title: Experience of the Nationwide Gambling Self-exclusion Service Spelpaus - Effects and Limitations of a Unique Harm Reduction Instrument for Problem Gambling
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Principal Investigator, Anders C Håkansson, Consultant physician, professor, Region Skane
Other Study IDs: Spelpaus study
Record Dates: First submitted 2022-12-27; First posted 2023-01-20 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Gambling Disorder; Problem Gambling
Keywords: gambling disorder; problem gambling; concerned significant others; self-exclusion; harm reduction
MeSH Terms: conditions — Gambling; Harm Reduction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals with a gambling problem: Recruited from a gambling disorder treatment unit and/or from social media advertising addressing individuals with a gambling problem.
  Interventions: Behavioral: Voluntary self-exclusion from gambling ('Spelpaus')
- Concerned significant others: Recruited as concerned signifiant others of patients at a gambling disorder treatment unit and/or in social media advertising addressing concerned significant others of individuals with a gambling problem.
  Interventions: Behavioral: Voluntary self-exclusion from gambling ('Spelpaus')

INTERVENTIONS:
Behavioral: Voluntary self-exclusion from gambling ('Spelpaus') — Voluntary self-exclusion from gambling, using the government-based, official service 'Spelpaus' (literally 'play break')

SUMMARY:
Qualitative interview study addressing the effects and limitations of a unique, government-based, nationwide self-exclusion service for the reduction of gambling-related harm. This service, which allows for individuals at risk of gambling problems (and for anyone) to self-exclude from all licensed gambling in the country, is unique in its nationwide, non-gambling-operator-dependent and multi-operator design. It is a promising tool for the prevention and harm reduction in relation to problem gambling and gambling disorder, but emerging research data report considerable limitations including high access to non-licensed gambling allowing users to breach the voluntary self-exclusion and relapse into hazardous gambling practices. This study will examine effects and limitations of the system, for gamblers and for concerned significant others of gamblers, through qualitative interviews addressing their experience of the system.

ELIGIBILITY:
Inclusion Criteria:

* Patient at a gambling disorder unit or self-recruited through social media advertising and defining as a person with a gambling problem, and/or concerned significant other of a patient at a gambling disorder unit or self-recruited through social media advertising and defining as a concerned significant other of a person with a gambling problem.

Exclusion Criteria:

* Inability to provide informed study consent and to carry out a qualitative research interview, due to language difficulties and/or cognitive problems.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 1. Patients at a gambling disorder unit, or self-recruited through social media advertising and defining as a person with a gambling problem
  2. Concerned significant others of patients at a gambling disorder unit or self-recruited through social media advertising and defining as a concerned significant other of a person with a gambling problem.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-02-13 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Qualitative reporting of self-perceived effects from self-exclusion | Since 2019
  Subjective perception of favorable effects on gambling behavior or well-being
Qualitative reporting of self-perceived harm or limitations from self-exclusion | Since 2019
  Subjective perception of negative impact or lack of improvement with respect to gambling behavior or well-being

CONTACTS AND LOCATIONS:
Overall Officials: Anders Håkansson, PhD, Principal Investigator — Region Skåne; Helena Hansson, PhD, Study Director — Lund University, School of Social Work
Locations (1):
- Malmö Addiction Center, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hakansson A, Tjernberg J, Hansson H. Effects and Limitations of a Unique, Nationwide, Self-Exclusion Service for Gambling Disorder and Its Self-Perceived Effects and Harms in Gamblers: Protocol for a Qualitative Interview Study. JMIR Res Protoc. 2023 Nov 14;12:e47528. doi: 10.2196/47528. PMID 37962917